CLINICAL TRIAL: NCT01956773
Title: Family Health History in Diverse Care Settings
Brief Title: Family Health History in Diverse Care Settings (FHH)
Acronym: FHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00043372; Pro00047666 (Other: DUHS IRB)
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Diabetes; Heart Disease; Cancer
Keywords: family health history; prevention; genetic risk; clinical decision support
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MeTree - Patient (Experimental): MeTree collects family health history data and generates risk scores and specific risk-based recommendation for preventive care to patients as clinical decision support.
  Interventions: Other: MeTree
- MeTree - Provider (Experimental): MeTree collects family health history data and generates risk scores and specific risk-based recommendation for preventive care to providers as clinical decision support.
  Interventions: Other: MeTree

INTERVENTIONS:
Other: MeTree — Software program collecting family health history and generating clinical decision support for risk-based preventive care

SUMMARY:
The outcome of this research will be a demonstration that family health history (FHH) risk data can be used efficiently to deliver more effective healthcare in geographically and ethnically diverse clinical care environments. Although FHH is a standard component of the medical interview its widespread adoption is hindered by three major barriers: (1) a dearth of standard collection methods; (2) the absence of health care provider access to complete FHH information; and (3) the need for clinical guidance for the interpretation and use of FHH. In addition, the time constraints of the busy provider and poor integration of FHH with paper medical records or electronic medical records (EMR) impede its widespread use. The investigators hypothesize that patient-driven and electronic collection of FHH for risk stratification will promote more informed decision-making by patients and providers, and improves adherence to risk-stratified preventive care guidelines. The study team will use an implementation sciences approach to integrate an innovative FHH system that collects FHH from patients. Intermountain Healthcare will provide the information technology expertise with EMR design to develop an innovative solution to a storage model standard for FHH data as well as a centralized standards-compliant open clinical decision support (OpenCDS) rule development architecture to analyze FHH and to generate evidence-based, individualized, disease risk, preventive care recommendations for both patients and providers.

DETAILED DESCRIPTION:
Five health care delivery organizations will participate in this demonstration project: Duke University, the Medical College of Wisconsin, the Air Force, Essentia Health, and the University of North Texas Health Science Center. The study will take place in 'real world' clinical, socio-cultural, and demographically diverse (rural, underserved, academic, family medicine) care clinics (n=34) in 5 states (CA, MN, NC, WI, TX) that include genomic medicine 'early adopter' and 'naïve' sites, as well as those that are EMR-enabled and others that are not. The study team will recruit a minimum of 7000 English or Spanish speaking adults over a 3-year period and will capture process metrics and outcomes that are measured in the course of usual care. The goals are: 1) To optimize the collection of patient entered FHH in diverse clinical environments for coronary heart disease, thrombosis, and selected cancers, 2) to export FHH data to an OpenCDS platform and return CDS results to providers and patients (and to EMRs where relevant) and to explore the integration of genetic risk and FHH data at selected sites, 3) to assess the clinical and personal utility of FHH using a pragmatic observational study design to assess reach, adoption, integrity, exposure, and sustainability, and to capture, analyze, and report effectiveness outcomes at each stakeholder level: patient, provider, and clinic/system, and 4) to take a leadership role in the dissemination of guidelines for FHH intervention across in diverse practice settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age
* Scheduled for a well visit appointment in selected clinics
* English and Spanish speaking
* Able to provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2620 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey S Ginsburg, MD PHD, Principal Investigator — Duke University, Institute for Genome Science and Policy; Lori Orlando, MD, Principal Investigator — Duke University, Department of Medicine
Locations (5):
- United States (5):
  - David Grant Medical Center, Fairfield, California
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Wu RR, Myers RA, Neuner J, McCarty C, Haller IV, Harry M, Fulda KG, Dimmock D, Rakhra-Burris T, Buchanan A, Ginsburg GS, Orlando LA. Implementation-effectiveness trial of systematic family health history based risk assessment and impact on clinical disease prevention and surveillance activities. BMC Health Serv Res. 2022 Dec 6;22(1):1486. doi: 10.1186/s12913-022-08879-2. PMID 36474257
- [Derived] Orlando LA, Wu RR, Myers RA, Neuner J, McCarty C, Haller IV, Harry M, Fulda KG, Dimmock D, Rakhra-Burris T, Buchanan A, Ginsburg GS. At the intersection of precision medicine and population health: an implementation-effectiveness study of family health history based systematic risk assessment in primary care. BMC Health Serv Res. 2020 Nov 7;20(1):1015. doi: 10.1186/s12913-020-05868-1. PMID 33160339
- [Derived] Wu RR, Myers RA, Buchanan AH, Dimmock D, Fulda KG, Haller IV, Haga SB, Harry ML, McCarty C, Neuner J, Rakhra-Burris T, Sperber N, Voils CI, Ginsburg GS, Orlando LA. Effect of Sociodemographic Factors on Uptake of a Patient-Facing Information Technology Family Health History Risk Assessment Platform. Appl Clin Inform. 2019 Mar;10(2):180-188. doi: 10.1055/s-0039-1679926. Epub 2019 Mar 13. PMID 30866001
- [Derived] Wu RR, Myers RA, McCarty CA, Dimmock D, Farrell M, Cross D, Chinevere TD, Ginsburg GS, Orlando LA; Family Health History Network. Protocol for the "Implementation, adoption, and utility of family history in diverse care settings" study. Implement Sci. 2015 Nov 24;10:163. doi: 10.1186/s13012-015-0352-8. PMID 26597091

RESULTS

PARTICIPANT FLOW:
Groups:
- MeTree - Patients: MeTree collects family health history data and generates risk scores and specific risk-based recommendation for preventive care to patients and providers as clinical decision support.
  MeTree: Software program collecting family health history and generating clinical decision support for risk-based preventive care
- MeTree - Providers: Providers using MeTree risk assessment program for clinical decision support
Period: Overall Study
Arm/Group | MeTree - Patients | MeTree - Providers
Started | 2520 | 100
Completed | 1892 | 99
Not Completed | 628 | 1
Not completed — Lost to Follow-up | 628 | 1

BASELINE CHARACTERISTICS:
Groups:
- MeTree - Patients: MeTree collects family health history data and generates risk scores and specific risk-based recommendation for preventive care to patients as clinical decision support.
  MeTree: Software program collecting family health history and generating clinical decision support for risk-based preventive care
- MeTree - Providers: MeTree collects family health history data and generates risk scores and specific risk-based recommendation for preventive care to Providers as clinical decision support.
  MeTree: Software program collecting family health history and generating clinical decision support for risk-based preventive care
- Total: Total of all reporting groups
Arm/Group | MeTree - Patients | MeTree - Providers | Total
Number analyzed (Participants) | 2520 | 100 | 2620
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1666 | 99 | 1765
  >=65 years | 854 | 1 | 855
Age, Continuous [Median (Full Range); unit: years] | 59 [19 to 94] | 41 [26 to 66] | 59 [19 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1725 | 61 | 1786
  Male | 795 | 39 | 834
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 0 | 42
  Not Hispanic or Latino | 1578 | 0 | 1578
  Unknown or Not Reported | 900 | 100 | 1000
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 30 | 12 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 165 | 1 | 166
  White | 1779 | 81 | 1860
  More than one race | 48 | 1 | 49
  Unknown or Not Reported | 495 | 3 | 498
Region of Enrollment [Number; unit: participants]
  United States | 2520 | 100 | 2620

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Uptake of Genetic Counseling for Those at Risk of Hereditary Conditions at 1 Year
Description: How many patients identified as meeting criteria for genetic counseling, how many providers ordered genetic counseling, and how many patients adhere to the provider recommendation at 1 year.
Time Frame: Baseline, 3 and 12 months
Population: Patients who completed intervention and meeting criteria for genetic counseling
Measure: Count of Participants; unit: Participants
Arm/Group | MeTree - Patients
Number analyzed (Participants) | 1838
Participants
  Patients who met genetic counseling criteria | 571
  Patients who received Genetic Counseling Order: number analyzed (Participants) | 571
  Patients who received Genetic Counseling Order | 49
  Patients adhered to provider's recommendation-1yr: number analyzed (Participants) | 49
  Patients adhered to provider's recommendation-1yr | 32
  Providers who placed Genetic counseling order: number analyzed (Participants) | 77
  Providers who placed Genetic counseling order | 31

2. Secondary Outcome: Number of Participants Reporting Satisfaction When Using the MeTree Tool
Description: The study will assess satisfaction associated with using the MeTree tool via 3 months survey after completing the family health history collection. The participant were asked their level of satisfaction with their experience using the web-based portal to enter information for their provider before their appointment
Time Frame: 3 months
Population: Patients who completed 3 months post survey and reported their level of satisfaction
Measure: Count of Participants; unit: Participants
Arm/Group | MeTree - Patients
Number analyzed (Participants) | 1102
Participants
  Superior | 69
  Above Average | 459
  Very Satisfactory | 474
  Somewhat unsatisfactory | 59
  Very Poor | 23
  Not Answered | 18

3. Secondary Outcome: Number of Participants Reporting Comfort When Using the MeTree Tool
Description: The study will assess comfort associated with using the MeTree tool via 3 months survey after completing the family health history collection. The participant were asked if the MeTree program was easy to use
Time Frame: 3 months
Population: Patients who completed 3 months post survey and reported on their level of comfort
Measure: Count of Participants; unit: Participants
Arm/Group | MeTree - Patients
Number analyzed (Participants) | 1102
Participants
  Do not know | 20
  No | 78
  Yes | 988
  did not answer | 16

4. Secondary Outcome: Number of Participants Reporting Anxiety When Using the MeTree Tool
Description: The study will assess anxiety associated with using the MeTree tool via 3 months survey after completing the family health history collection. The participant were asked if answering the questions made them anxious
Time Frame: 3 months
Population: Patients who completed 3 months post survey and reported on anxiety with answering the questions
Measure: Count of Participants; unit: Participants
Arm/Group | MeTree - Patients
Number analyzed (Participants) | 1102
Participants
  Do not know | 14
  No | 1032
  Yes | 43
  Did not answer | 13

5. Secondary Outcome: Number of Participants Reporting Preparedness When Using the MeTree Tool
Description: The study will assess preparedness associated with using the MeTree tool via 3 months survey after completing the family health history collection. The participants were asked if they had enough information about some people in their family when completing MeTree
Time Frame: 3 months
Population: Patients who completed 3 months post survey and reported on preparedness
Measure: Count of Participants; unit: Participants
Arm/Group | MeTree - Patients
Number analyzed (Participants) | 1102
Participants
  Do not know | 59
  No | 377
  Yes | 646
  Did not answer | 20

6. Secondary Outcome: Number of Physicians Who Gave Their Perceptions of Satisfaction and the MeTree Tool's Impact on Work Load
Description: Evaluate physicians' perceptions of satisfaction, the MeTree tool's impact on work load and its effectiveness via survey and informal interviews at 3 months.
Time Frame: 3 months
Population: Consented providers who completed provider post implementation survey
Measure: Count of Participants; unit: Participants
Arm/Group | MeTree - Providers
Number analyzed (Participants) | 43
Participants
  Acceptable Tool - Yes | 34
  Acceptable Tool - No | 9

7. Secondary Outcome: Number of Providers Who Were Successfully Using MeTree in Their Clinical Work Flow
Description: Evaluate which providers were successfully using MeTree in their clinical work flow and which patients are successfully using MeTree for their care. (surveys, monitoring of clinical workflow, patient recruitment reflects underlying clinic population)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | MeTree - Providers
Number analyzed (Participants) | 100
Participants | 100

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-Cause Mortality and Serious Adverse Events were not monitored/assessed for either Arm/Group
Arm/Group | MeTree - Patients | MeTree - Providers
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2520 | 0/100

LIMITATIONS AND CAVEATS:
12 mo survey ended early w/ approved by Duke IRB. Sufficient data obtained to perform the scientific analysis; the overall status of the study is still active, not recruiting. Participant contact completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT01956773/Prot_SAP_000.pdf